CLINICAL TRIAL: NCT00338247
Title: An Open-Label Expanded Access Study of Lapatinib and Capecitabine Therapy in Subjects With ErbB2 Overexpressing Locally Advanced or Metastatic Breast Cancer
Brief Title: EAP (Expanded Access Protocol) Of Lapatinib Combined With Capecitabine In Metastatic Breast Cancer
Status: Approved for marketing | Type: Expanded Access
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: EGF103659
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Neoplasms, Breast
Keywords: advanced; TYKERB; HER2 positive; Stage IIIc; ErbB2 positive; GW572016; metastatic; Stage IIIb; breast cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Lapatinib; Capecitabine

INTERVENTIONS:
Drug: lapatinib + capecitabine — Experimental

SUMMARY:
This study will provide pre-approval drug access to lapatinib, in combination with capecitabine, to patients whose breast cancer had progressed on other therapies

ELIGIBILITY:
Inclusion criteria:

* May have received prior lapatinib in another trial. Previous capecitabine (as previous agent or non-lapatinib containing regimen) is also permitted.
* Prior treatment with hormonal therapy is allowed.
* Must have advanced or metastatic breast cancer with progression (as assessed by modified RECIST) after prior therapy, which must include all of the following: prior treatment with an anthracycline, a taxane, and trastuzumab alone or in combination with other therapy. Trastuzumab must have been administered in the adjuvant, or locally advanced or metastatic setting.
* Must have tumors that overexpress ErbB2 defined as +3 by IHC or FISH positive for ErbB2 gene amplification. The status of ErbB2 expression must be documented prior to study entry.
* Must be >/= 18 years of age
* Life expectancy of > 8 weeks
* Must have recovered from side effects of previous treatment
* Patients with CNS mets are eligible provided treatment with prohibited medications as listed in the protocol are not required
* Cardiac ejection fraction must be within the institutional range of normal as measured by ECHO. MUGA scans are allowed if ECHOs cannot be performed
* Able to swallow and retain oral medications
* Must have adequate hematologic, hepatic and renal function

Exclusion criteria:

* Pregnant or lactating females
* Malabsorption syndrome, disease significantly affecting GI function, or resection of the stomach or bowel, or ulcerative colitis
* Concurrent disease or condition that would make the patient inappropriate for study participation
* Unresolved or unstable toxicity from prior administration of another investigational drug and/or prior cancer treatment
* Uncontrolled infection
* Active cardiac disease defined as history of uncontrolled or symptomatic angina; history of arrhythmias requiring medication, or clinically significant, with the exception of asymptomatic atrial fibrillation requiring anticoagulation; MI < 6 months from study entry; uncontrolled or symptomatic CHF; ejection fraction below the institutional normal limit; any other cardiac condition that would make this protocol unreasonably hazardous for the patient
* Receiving concurrent chemotherapy (other than capecitabine), radiation therapy, immunotherapy, biologic therapy or hormonal therapy for cancer. Concurrent therapy with bisphosphonates is allowed
* History of allergic reaction attributed to compounds of similar composition to lapatinib or any excipients
* History of allergic reactions attributed to compounds of similar chemical composition to capecitabine, fluorouracil or excipients
* Known DPD deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (392):
- United States (138):
  - Novartis Investigative Site, Huntsville, Alabama
  - Novartis Investigative Site, Anchorage, Alaska
  - Novartis Investigative Site, Glendale, Arizona
  - Novartis Investigative Site, Fayetteville, Arkansas
  - Novartis Investigative Site, Little Rock, Arkansas
  - Novartis Investigative Site, Bellflower, California
  - Novartis Investigative Site, Burbank, California
  - Novartis Investigative Site, Gilroy, California
  - Novartis Investigative Site, Long Beach, California
  - Novartis Investigative Site, Newport Beach, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Santa Rosa, California
  - Novartis Investigative Site, Stockton, California
  - Novartis Investigative Site, Aurora, Colorado
  - Novartis Investigative Site, Boulder, Colorado
  - Novartis Investigative Site, Lafayette, Colorado
  - Novartis Investigative Site, Hartford, Connecticut
  - Novartis Investigative Site, Manchester, Connecticut
  - Novartis Investigative Site, New Havey, Connecticut
  - Novartis Investigative Site, Norwich, Connecticut
  - Novartis Investigative Site, Washington D.C., District of Columbia
  - Novartis Investigative Site, Fort Lauderdale, Florida
  - Novartis Investigative Site, Fort Myers, Florida
  - Novartis Investigative Site, Fort Walton Beach, Florida
  - Novartis Investigative Site, Gainesville, Florida
  - Novartis Investigative Site, Hollywood, Florida
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Augusta, Georgia
  - Novartis Investigative Site, Brunswick, Georgia
  - Novartis Investigative Site, Macon, Georgia
  - Novartis Investigative Site, Marietta, Georgia
  - Novartis Investigative Site, Tucker, Georgia
  - Novartis Investigative Site, Honolulu, Hawaii
  - Novartis Investigative Site, Boise, Idaho
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Decatur, Illinois
  - Novartis Investigative Site, Galesburg, Illinois
  - Novartis Investigative Site, Highland Park, Illinois
  - Novartis Investigative Site, Joliet, Illinois
  - Novartis Investigative Site, Peoria, Illinois
  - Novartis Investigative Site, Zion, Illinois
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Bettendorf, Iowa
  - Novartis Investigative Site, Cedar Rapids, Iowa
  - Novartis Investigative Site, Council Bluffs, Iowa
  - Novartis Investigative Site, Sioux City, Iowa
  - Novartis Investigative Site, Waterloo, Iowa
  - Novartis Investigative Site, Baton Rouge, Louisiana
  - Novartis Investigative Site, Metairie, Louisiana
  - Novartis Investigative Site, Portland, Maine
  - Novartis Investigative Site, Scarborough, Maine
  - Novartis Investigative Site, Waterville, Maine
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Chevy Chase, Maryland
  - Novartis Investigative Site, Frederick, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Fall River, Massachusetts
  - Novartis Investigative Site, Peabody, Massachusetts
  - Novartis Investigative Site, Ann Arbor, Michigan
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Royal Oak, Michigan
  - Novartis Investigative Site, Troy, Michigan
  - Novartis Investigative Site, Duluth, Minnesota
  - Novartis Investigative Site, Jackson, Mississippi
  - Novartis Investigative Site, Columbia, Missouri
  - Novartis Investigative Site, Kalamazoo, Missouri
  - Novartis Investigative Site, Kansas City, Missouri
  - Novartis Investigative Site, Springfield, Missouri
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Billings, Montana
  - Novartis Investigative Site, Great Falls, Montana
  - Novartis Investigative Site, Grand Island, Nebraska
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, North Platte, Nebraska
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Exeter, New Hampshire
  - Novartis Investigative Site, Flemington, New Jersey
  - Novartis Investigative Site, Freehold, New Jersey
  - Novartis Investigative Site, Little Silver, New Jersey
  - Novartis Investigative Site, Livingston, New Jersey
  - Novartis Investigative Site, Mountain Lakes, New Jersey
  - Novartis Investigative Site, Newark, New Jersey
  - Novartis Investigative Site, Buffalo, New York
  - Novartis Investigative Site, East Setauket, New York
  - Novartis Investigative Site, East Syracuse, New York
  - Novartis Investigative Site, Fresh Meadows, New York
  - Novartis Investigative Site, Glens Falls, New York
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Asheville, North Carolina
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Fayetteville, North Carolina
  - Novartis Investigative Site, Greensboro, North Carolina
  - Novartis Investigative Site, Bismarck, North Dakota
  - Novartis Investigative Site, Fargo, North Dakota
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Sandusky, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Tulsa, Oklahoma
  - Novartis Investigative Site, Klamath Falls, Oregon
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Drexel Hill, Pennsylvania
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Pottstown, Pennsylvania
  - Novartis Investigative Site, Sayre, Pennsylvania
  - Novartis Investigative Site, State College, Pennsylvania
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Columbia, South Carolina
  - Novartis Investigative Site, Florence, South Carolina
  - Novartis Investigative Site, Mt. Pleasant, South Carolina
  - Novartis Investigative Site, Knoxville, Tennessee
  - Novartis Investigative Site, Memphis, Tennessee
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Arlington, Texas
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, El Paso, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Salt Lake City, Utah
  - Novartis Investigative Site, Fairfax, Virginia
  - Novartis Investigative Site, Richmond, Virginia
  - Novartis Investigative Site, Kennewick, Washington
  - Novartis Investigative Site, Mount Vernon, Washington
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Tacoma, Washington
  - Novartis Investigative Site, Walla Walla, Washington
  - Novartis Investigative Site, Morgantown, West Virginia
  - Novartis Investigative Site, Green Bay, Wisconsin
  - Novartis Investigative Site, La Crosse, Wisconsin
  - Novartis Investigative Site, Marshfield, Wisconsin
- Australia (15):
  - Novartis Investigative Site, Kogarah, New South Wales
  - Novartis Investigative Site, North Sydney, New South Wales
  - Novartis Investigative Site, Port Macquarie, New South Wales
  - Novartis Investigative Site, Waratah, New South Wales
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Herston, Queensland
  - Novartis Investigative Site, South Brisbane, Queensland
  - Novartis Investigative Site, Bedford Park, South Australia
  - Novartis Investigative Site, Hobart, Tasmania
  - Novartis Investigative Site, Box Hill, Victoria
  - Novartis Investigative Site, Fitzroy, Victoria
  - Novartis Investigative Site, Geelong, Victoria
  - Novartis Investigative Site, Wodonga, Victoria
  - Novartis Investigative Site, Nedlands, Western Australia
  - Novartis Investigative Site, Perth, Western Australia
- Austria (5):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Innsbruck
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Belgium (9):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Charleroi
  - Novartis Investigative Site, Edegem
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Haine-Saint-Paul
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Wilrijk
  - Novartis Investigative Site, Yvoir
- Brazil (5):
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Jaú, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Novartis Investigative Site, Sofia, Bulgaria
- Canada (7):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Winnipeg, Manitoba
  - Novartis Investigative Site, Moncton, New Brunswick
  - Novartis Investigative Site, Greater Sudbury, Ontario
  - Novartis Investigative Site, Oshawa, Ontario
  - Novartis Investigative Site, Greenfield Park, Quebec
  - Novartis Investigative Site, Saskatoon, Saskatchewan
- Novartis Investigative Site, Santiago, Región Metro de Santiago, Chile
- China (8):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Dalian, Liaoning
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
- Novartis Investigative Site, Stróvolos, Cyprus
- Czechia (3):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Prague
- Denmark (5):
  - Novartis Investigative Site, Århus C
  - Novartis Investigative Site, Copenhagen
  - Novartis Investigative Site, Odense C
  - Novartis Investigative Site, Roskilde
  - Novartis Investigative Site, Vejle
- Estonia (2):
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- Finland (5):
  - Novartis Investigative Site, Hämeenlinna
  - Novartis Investigative Site, Helsinki
  - Novartis Investigative Site, Kangasala
  - Novartis Investigative Site, Kuopio
  - Novartis Investigative Site, OYS
- Germany (21):
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Stuttgart, Baden-Wurttemberg
  - Novartis Investigative Site, Tübingen, Baden-Wurttemberg
  - Novartis Investigative Site, Augsburg, Bavaria
  - Novartis Investigative Site, Hamburg, Hamburg
  - Novartis Investigative Site, Marburg, Hesse
  - Novartis Investigative Site, Wiesbaden, Hesse
  - Novartis Investigative Site, Braunschweig, Lower Saxony
  - Novartis Investigative Site, Hanover, Lower Saxony
  - Novartis Investigative Site, Bonn, North Rhine-Westphalia
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Düsseldorf, North Rhine-Westphalia
  - Novartis Investigative Site, Ibbenbueren, North Rhine-Westphalia
  - Novartis Investigative Site, Mönchengladbach, North Rhine-Westphalia
  - Novartis Investigative Site, Troisdorf, North Rhine-Westphalia
  - Novartis Investigative Site, Mainz, Rhineland-Palatinate
  - Novartis Investigative Site, Saarbrücken, Saarland
  - Novartis Investigative Site, Halle, Saxony-Anhalt
  - Novartis Investigative Site, Magdeburg, Saxony-Anhalt
  - Novartis Investigative Site, Lübeck, Schleswig-Holstein
  - Novartis Investigative Site, Berlin, State of Berlin
- Greece (3):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Heraklion, Crete
  - Novartis Investigative Site, Marousi
- Hong Kong (2):
  - Novartis Investigative Site, Pokfulam
  - Novartis Investigative Site, Shatin
- Novartis Investigative Site, Reykjavik, Iceland
- Novartis Investigative Site, Jakarta, Indonesia
- Ireland (4):
  - Novartis Investigative Site, Dublin
  - Novartis Investigative Site, Galway
  - Novartis Investigative Site, Tallaght, Dublin
  - Novartis Investigative Site, Wilton, Cork
- Israel (7):
  - Novartis Investigative Site, Beersheba
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Rehovot
  - Novartis Investigative Site, Tel Aviv
- Italy (25):
  - Novartis Investigative Site, Bari, Apulia
  - Novartis Investigative Site, San Giovanni Rotondo (FG), Apulia
  - Novartis Investigative Site, Potenza, Basilicate
  - Novartis Investigative Site, Reggio Calabria, Calabria
  - Novartis Investigative Site, Napoli, Campania
  - Novartis Investigative Site, Forlì, Emilia-Romagna
  - Novartis Investigative Site, Modena, Emilia-Romagna
  - Novartis Investigative Site, Aviano (PN), Friuli Venezia Giulia
  - Novartis Investigative Site, Rome, Lazio
  - Novartis Investigative Site, Genoa, Liguria
  - Novartis Investigative Site, Bergamo, Lombardy
  - Novartis Investigative Site, Milan, Lombardy
  - Novartis Investigative Site, Candiolo (TO), Piedmont
  - Novartis Investigative Site, Turin, Piedmont
  - Novartis Investigative Site, Palermo, Sicily
  - Novartis Investigative Site, Bolzano, Trentino-Alto Adige
  - Novartis Investigative Site, Florence, Tuscany
  - Novartis Investigative Site, Pisa, Tuscany
  - Novartis Investigative Site, Perugia, Umbria
  - Novartis Investigative Site, Ancona
  - Novartis Investigative Site, Cagliari
  - Novartis Investigative Site, Chieti
  - Novartis Investigative Site, Macerata
  - Novartis Investigative Site, Padua
  - Novartis Investigative Site, Trieste
- Novartis Investigative Site, Luxembourg, Luxembourg
- Malaysia (2):
  - Novartis Investigative Site, Kuala Lumpur
  - Novartis Investigative Site, Petaling Jaya Selangor
- Novartis Investigative Site, Floriana, Malta
- Mexico (5):
  - Novartis Investigative Site, Tijuana, Baja California Norte
  - Novartis Investigative Site, Toluca, Edo Mex, State of Mexico
  - Novartis Investigative Site, Mérida, Yucatán
  - Novartis Investigative Site, Durango
  - Novartis Investigative Site, Mexico City
- Netherlands (8):
  - Novartis Investigative Site, Amersfoort
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Dordrecht
  - Novartis Investigative Site, Enschede
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Leeuwarden
  - Novartis Investigative Site, Leiden
  - Novartis Investigative Site, Maastricht
- New Zealand (3):
  - Novartis Investigative Site, Christchurch
  - Novartis Investigative Site, Dunedin
  - Novartis Investigative Site, Newtown, Wellington
- Novartis Investigative Site, Lima, Lima Province, Peru
- Philippines (4):
  - Novartis Investigative Site, Makati City
  - Novartis Investigative Site, Pasay
  - Novartis Investigative Site, Quezon City
  - Novartis Investigative Site, Sampaloc Manila
- Poland (8):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Bydgoszcz
  - Novartis Investigative Site, Elblag
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Gliwice
  - Novartis Investigative Site, Olsztyn
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Warsaw
- Portugal (3):
  - Novartis Investigative Site, Evora
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
- Romania (4):
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Iași
  - Novartis Investigative Site, Sibiu
  - Novartis Investigative Site, Timișoara
- Russia (3):
  - Novartis Investigative Site, Irkutsk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Nizhny Novgorod
- Novartis Investigative Site, Singapore, Singapore
- Slovakia (4):
  - Novartis Investigative Site, Banská Bystrica
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Poprad
- Slovenia (2):
  - Novartis Investigative Site, Ljubljana
  - Novartis Investigative Site, Maribor
- South Korea (5):
  - Novartis Investigative Site, Kyunggi-do
  - Novartis Investigative Site, Pusan
  - Novartis Investigative Site, Seodaemun-gu, Seoul
  - Novartis Investigative Site, Seoul
  - Novartis Investigative Site, Songpa-gu, Seoul
- Spain (21):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Basurto/Bilbao
  - Novartis Investigative Site, Burgos
  - Novartis Investigative Site, Cáceres
  - Novartis Investigative Site, Elche
  - Novartis Investigative Site, Girona
  - Novartis Investigative Site, Jaén
  - Novartis Investigative Site, Lleida
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Murcia
  - Novartis Investigative Site, Palencia
  - Novartis Investigative Site, Palma de Mallorca
  - Novartis Investigative Site, Pamplona
  - Novartis Investigative Site, Pontevedra
  - Novartis Investigative Site, San Sebastián
  - Novartis Investigative Site, Santa Cruz de Tenerife
  - Novartis Investigative Site, Santiago
  - Novartis Investigative Site, Toledo
  - Novartis Investigative Site, Valencia
  - Novartis Investigative Site, Zaragoza
- Sweden (5):
  - Novartis Investigative Site, Jönköping
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Umeå
  - Novartis Investigative Site, Uppsala
- Switzerland (8):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Chur
  - Novartis Investigative Site, Geneva
  - Novartis Investigative Site, Mendrisio
  - Novartis Investigative Site, Neuchâtel
  - Novartis Investigative Site, Sankt Gallen
  - Novartis Investigative Site, Zurich
- Taiwan (5):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Tainan County
  - Novartis Investigative Site, Taipei
- Thailand (3):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
  - Novartis Investigative Site, Pathum Thani
- Ukraine (4):
  - Novartis Investigative Site, Chernivtsi
  - Novartis Investigative Site, Kiev
  - Novartis Investigative Site, Odesa
  - Novartis Investigative Site, Rivne
- United Kingdom (22):
  - Novartis Investigative Site, Cambridge, Cambridgeshire
  - Novartis Investigative Site, Chelmsford, Essex
  - Novartis Investigative Site, Northwood, Middlesex
  - Novartis Investigative Site, Edinburgh, Midlothian
  - Novartis Investigative Site, Belfast
  - Novartis Investigative Site, Bournemouth
  - Novartis Investigative Site, Brighton
  - Novartis Investigative Site, Bristol
  - Novartis Investigative Site, Cardiff
  - Novartis Investigative Site, Cheltenham
  - Novartis Investigative Site, Colchester
  - Novartis Investigative Site, Cumbria
  - Novartis Investigative Site, Denbighshire
  - Novartis Investigative Site, Hartshill, Stoke-on-Trent
  - Novartis Investigative Site, Lindley, Huddersfield
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Nottingham
  - Novartis Investigative Site, Peterborough
  - Novartis Investigative Site, Poole, Dorset
  - Novartis Investigative Site, Portsmouth
  - Novartis Investigative Site, Shrewsbury

REFERENCES:
- [Derived] Ro J, Park S, Kim S, Kim TY, Im YH, Rha SY, Chung JS, Moon H, Santillana S. Clinical outcomes of HER2-positive metastatic breast cancer patients with brain metastasis treated with lapatinib and capecitabine: an open-label expanded access study in Korea. BMC Cancer. 2012 Jul 28;12:322. doi: 10.1186/1471-2407-12-322. PMID 22839200
- [Derived] Wang L, Zhang Q, Zhang J, Sun S, Guo H, Jia Z, Wang B, Shao Z, Wang Z, Hu X. PI3K pathway activation results in low efficacy of both trastuzumab and lapatinib. BMC Cancer. 2011 Jun 15;11:248. doi: 10.1186/1471-2407-11-248. PMID 21676217